CLINICAL TRIAL: NCT07220772
Title: An Open-Label Study of Mibavademab (REGN4461), a Leptin Receptor Agonist, for the Treatment of Monogenic Obesity Due to Biallelic Loss of Function Variants of the LEP Gene
Brief Title: A Study Evaluating Mibavademab Treatment of Obesity Due to Leptin (LEP) Gene Mutations in Children, Adolescents and Adults
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R4461-MOB-2471; 2024-518674-14-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2025-10-22; First posted 2025-10-24 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Monogenic Obesity
Keywords: Biallelic loss of function variants of the LEP gene mutations; Leptin deficiency
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Mibavademab (Experimental)
  Interventions: Drug: Mibavademab

INTERVENTIONS:
Drug: Mibavademab — Administered as per the protocol
  Other Names: REGN4461

SUMMARY:
This study is researching an experimental drug called mibavademab. The study is focused on patients with a condition called monogenic obesity. Monogenic obesity is caused by a change in the leptin gene that keeps it from working properly. This causes the body to not be able to feel full or control feelings of hunger.

The aim of the study is to see how well mibavademab controls the body weight and how safe it is.

The study is looking at several other research questions, including:

* How much mibavademab is in the blood at different times
* Whether the body makes proteins called antibodies against mibavademab (which could stop mibavademab from working as well or could lead to side effects)
* What side effects may happen from taking mibavademab

ELIGIBILITY:
Key Inclusion Criteria:

1. Has documented medical history of biallelic loss of function variants of the LEP gene prior to the screening visit
2. Has class ≥2 obesity at screening and at baseline, as defined in the protocol

Key Exclusion Criteria:

1. Unwilling or unable to provide, or have the treating physician provide, documented historical weight for at least 6 months prior to screening
2. History of bariatric surgery within approximately the past 12 months of study screening
3. History of weight loss of ≥5% of body weight in approximately the past 3 months of study screening
4. History of genetic causes of obesity other than/in addition to biallelic loss of function variants of the LEP gene
5. History of schizophrenia, bipolar disorder, or other mental illness that, in the opinion of the investigator, might pose a safety risk to participation in a clinical study of an investigational drug
6. Any suicidal ideation of type 4 or 5 on the Columbia Suicide Severity Rating Scale (C-SSRS) during screening or baseline, or any lifetime history of a suicide attempt, or any lifetime history of suicidal behavior, including ideation
7. Treatment with medications for weight loss or medications with known side effects of weight loss within the past approximately 3 months of study screening
8. Participants currently being treated with metreleptin, or a history of prior treatment with metreleptin as defined in the protocol

NOTE: Other Protocol-defined Inclusion/Exclusion Criteria Apply

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2025-12-19 (Estimated); Primary Completion 2027-04-09 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
Percent change in Body Mass Index (BMI) | Baseline to Week 24

SECONDARY OUTCOMES:
Percent change in BMI | Baseline to Week 52
Absolute change in BMI | Baseline, Through Week 52
Percent change in body weight | Baseline, Through Week 52
Absolute change in body weight | Baseline, Through Week 52
Change in waist circumference | Baseline, Through Week 52
  Participants aged ≥18 years
Change in absolute total fat mass by whole body DXA | Baseline, Through Week 52
Change in percent total fat mass by whole body DXA | Baseline, Through Week 52
Change in absolute regional fat mass by whole body DXA | Baseline, Through Week 52
Change in percent regional fat mass by whole body DXA | Baseline, Through Week 52
Change in scores in the symptoms of hyperphagia questionnaire | Baseline, Through Week 52
  Symptoms of Hyperphagia - Caregiver Version© is completed by a caregiver. Symptoms of Hyperphagia - Patient Version© is completed by the participants who are aged <12 years or for participants who are unable to self-complete. The questionnaires both assesses the frequency of hunger symptoms on a categorical scale (Never, 1 or 2 times, 3 or more times) over the past 24 hours and are scored combining the total scores across the items. Higher scores indicate greater severity.
Change in scores in the impacts of hyperphagia questionnaire | Baseline, Through Week 52
  For participants who are aged <12 years or for participants who are unable to self-complete, the Impacts of Hyperphagia - Caregiver Version© is completed by a caregiver. For participants aged ≥12 years who are able to self-report, the Impacts of Hyperphagia - Patient Version© is completed by the participant. Both questionnaires assess the impact of hyperphagia on a categorical scale (range: not at all, a little, moderately, a great deal). The participant version is scored using a total score across the 5 items. The caregiver version is scored separately for each section. Higher scores indicate a greater impact of hyperphagia.
Change in scores in the hunger questionnaire | Baseline, Through Week 52
  The Daily Hunger Assessment is a daily, single item measuring hunger for participants aged ≥12 years who are able to self-complete, participants are asked to rate their highest level of hunger over for the day, where "0" is "not hungry at all" to "10" the hungriest possible."
Number of treatment-emergent adverse events (TEAEs) | Through Week 65
Severity of TEAEs | Through Week 65
Concentrations of total mibavademab in serum | Through Week 65
Incidence of anti-drug antibody (ADA) to mibavademab | Through Week 65
Titer of ADA to mibavademab | Through Week 65

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/